CLINICAL TRIAL: NCT04974034
Title: Movement Disorders Analysis Using a Deep Learning Approach
Status: Completed | Type: Observational
Sponsor: Hospital Avicenne (Other)
Responsible Party: Principal Investigator, Desjardins Clement, Neurology Resident, Hospital Avicenne
Other Study IDs: CLEA-2019-83
Record Dates: First submitted 2021-07-03; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Bradykinesia; Parkinson Disease; Hypokinesia; Akinesia; Parkinsonian Syndrome; Parkinsonian Disorders
Keywords: Deep Learning; Bradykinesia; Parkinson Disease
MeSH Terms: conditions — Hypokinesia; Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bradykinesia is a key parkinsonian feature yet subjectively assessed by the MDS-UPDRS score, making reproducible measurements and follow-up challenging.

In a Movement Disorder Unit, the investigators acquired a large database of videos showing parkinsonian patients performing Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III protocols.

Using a Deep Learning approach on these videos, the investigators aimed to develop a tool to compute an objective score of bradykinesia from the three upper limb tests described in the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years

Exclusion Criteria:

* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients seen by a neurologist in the department of Neurology at Avicenne Hospital (Bobigny, France) between June 2019 and December 2020 were recorded during MDS-UPDRS examination.
  The investigators also included healthy volunteers on a voluntary basis.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III score | 1 day
  Automatic Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III for hand bradykinesia including the three following specific tasks (finger tapping, hand movements and pronation-supination movements of hand).
  The minimum score is 0. The maximum score is 12 Higher scores mean wors outcome

CONTACTS AND LOCATIONS:
Overall Officials: Clément Desjardins, MD, Principal Investigator — Hospital Avicenne; Bertrand Degos, MD,PhD, Study Director — Hospital Avicenne
Locations (1):
- Hospital Avicenne, Bobigny, Seine Saint Denis, France

IPD SHARING:
Plan to Share IPD: Undecided